CLINICAL TRIAL: NCT07353736
Title: Hemodynamic Mechanisms, Clinical Profiles, and Prognostic Factors in Patients With Cerebral Arteriovenous Malformations and Intracranial Aneurysms: An Observational Cohort Study
Brief Title: Cerebral Arteriovenous Malformation With Aneurysm: Epidemiology, Clinical Features, and Prognosis
Status: Not yet recruiting | Type: Observational
Sponsor: Duan Chuanzhi (Other)
Collaborators: Beijing Tiantan Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Shenzhen Second People's Hospital (Other); Guangdong 999 Brain Hospital (Other)
Responsible Party: Sponsor-Investigator, Duan Chuanzhi, Professor, Zhujiang Hospital
Organization: Zhujiang Hospital (Other)
Other Study IDs: LC2016ZD032
Record Dates: First submitted 2025-12-08; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-10

CONDITIONS: Cerebral Arteriovenous Malformation; Intracranial Arterial Diseases; Intra Cerebral Hemorrhage; Intracranial Aneurysm; Brain Diseases
Keywords: Hemodynamic Mechanisms; Prospective cohort study; Endovascular treatment; Cerebral Arteriovenous Malformation; Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Intracranial Arterial Diseases; Cerebral Hemorrhage; Intracranial Aneurysm; Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples from patients with different types of cerebral arteriovenous malformations combined with intracranial aneurysms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with cerebral arteriovenous malformations and intracranial aneurysms: Patients diagnosed with concomitant cerebral arteriovenous malformations and intracranial aneurysms by digital subtraction angiography (DSA), and/or magnetic resonance imaging (MRI), and/or computed tomographic angiography (CTA).

SUMMARY:
The study is a multicenter, prospective cohort study designed to assess the natural history, clinical safety and efficacy of various treatment strategies in patients with cerebral arteriovenous malformations (AVMs) and intracranial aneurysms.

DETAILED DESCRIPTION:
This study aims to evaluate the clinical safety and efficacy of different treatment strategies in patients with cerebral arteriovenous malformations (AVMs) combined with intracranial aneurysms (IAs) through a multicenter, large-sample, prospective observational cohort study. It will comprehensively analyze the epidemiological characteristics, clinical manifestations, associated risk factors, natural disease progression, and bleeding risks, as well as explore the hemodynamic mechanisms and genetic background differences. Clinical data, imaging findings, and blood samples will be collected from patients to investigate the impact of hemodynamics on aneurysm formation, rupture risk, and treatment outcomes. Additionally, the study will explore the genetic differences of AVM and IA patients and their correlation with clinical presentation and prognosis, ultimately providing a scientific basis for individualized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cerebral arteriovenous malformation and intracranial aneurysm confirmed by CTA, MRA, and/or DSA;
* Availability of complete clinical and imaging data;
* Provision of written informed consent by the patient or their legally authorized representative to participate in the study and undergo follow-up;
* Not concurrently participating in any other clinical trials that may interfere with the outcomes of this study.

Exclusion Criteria:

* Previous complete occlusion of the aneurysm and/or arteriovenous malformation prior to enrollment;
* Coexistence of other cerebrovascular diseases such as moyamoya disease, cerebral cavernous malformation, cerebral venous sinus thrombosis, etc.;
* Absence of DSA imaging data or poor image quality that precludes accurate evaluation of key anatomical and hemodynamic parameters of the AVM and intracranial aneurysm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated across eight neurosurgery centers who were confirmed by digital subtraction angiography (DSA), and/or magnetic resonance imaging (MRI), computed tomographic angiography (CTA) to have cerebral arteriovenous malformation and intracranial aneurysm.
Sampling Method: Non-Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Imaging Treatment Success Rate of Target Vascular Lesions | 3 months postoperatively, 6 months postoperatively, 1years postoperatively, and 2 years postoperatively
  his is a composite endpoint with stratified reporting by lesion type. It will separately calculate and report the success rates for the following two patient cohorts:
  For patients with intracranial aneurysms: Treatment success is defined as complete occlusion on postoperative digital subtraction angiography, assessed as Class I by the Raymond-Roy Occlusion Classification (RROC) or as Grade D by the O'Kelly-Marotta (OKM) grading scale.
  For patients with cerebral arteriovenous malformations (AVMs): Treatment success is defined as complete embolization on postoperative digital subtraction angiography, confirmed by the core laboratory or two independent assessors with no residual nidus opacification.
  Critical clarification: This composite measure does NOT calculate an overall arithmetic combined success rate. The final reported values will be two independent percentages.

SECONDARY OUTCOMES:
Incidence of perioperative complications | Perioperative period
  Perioperative complications include technical related complications (vascular rupture, thrombosis, etc.) and clinical complications (neurological deficits, infections, etc.)
Proportion of patients with hemorrhagic complications during follow-up period | within three years
  Including the type of bleeding (intracerebral hemorrhage/subarachnoid hemorrhage/intraventricular hemorrhage), specific location of bleeding,amount of bleeding;and determination of bleeding source: determine the source of bleeding from malformation or aneurysm through imaging examination.
Proportion of patients with poor functional prognosis | 3 months postoperatively, 6 months postoperatively,and one year postoperatively
  mRS score 3-6
Proportion of patients with good functional prognosis | 3 months postoperatively, 6 months postoperatively,and one year postoperatively
  mRS score 0-2

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, MD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No